CLINICAL TRIAL: NCT07248930
Title: An Observational Pilot Study Evaluating the Efficacy and Safety of LPS Adsorption Using the Efferon LPS NEO Device in Children With Thermal Burns
Brief Title: Lipopolysaccharide Adsorption (Efferon LPS NEO) in Children With Thermal Burns
Status: Recruiting | Type: Observational
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Other Study IDs: efferon-lps-2025-03
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Burns
Keywords: Hemoadsorption; Hemoperfusion; Extracorporeal therapy; LPS adsorption
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Baseline therapy + Efferon LPS NEO: Patients will receive standart therapy for thermal burns treatments and Efferon LPS NEO hemoadsorption procedure. Prospective enrollement.
  Interventions: Device: Efferon LPS NEO
- Control group: The retrospective control group will include patients from the same medical institution's records from the previous 3 years, matched to the study cohort using propensity score matching. These patients received standard therapy for thermal burns, which could include hemofiltration or hemodiafiltration procedures.

INTERVENTIONS:
Device: Efferon LPS NEO — Efferon LPS NEO, a medical device, which is a cylindrical body filled with a polymeric hemosorbent that selectively absorbs LPS and excess cytokines. Two hemoadsorption procedures will be performed per patient, with a duration of 6-12 hours each and an interval of 24-120 hours between procedures. The procedures may be administered in combination with hemofiltration or hemodiafiltration, as determined by the investigator.
  Groups: Baseline therapy + Efferon LPS NEO

SUMMARY:
This observational pilot study aims to identify criteria for evaluating the effectiveness of hemoadsorption with the Efferon LPS NEO device in pediatric burn injury. Participants will be prospectively assigned to the treatment group and compared with a retrospectively selected control group. Each patient in the treatment group will undergo two hemoadsorption sessions, each lasting 6-12 hours, with an interval of 24-120 hours between procedures. The sessions may be performed in combination with hemofiltration or hemodiafiltration at the discretion of the investigator.

DETAILED DESCRIPTION:
Extensive burns are a severe form of trauma that, according to the World Health Organization, cause more than 180,000 deaths worldwide each year. Despite advances in modern medicine, sepsis and other infectious complications remain the leading causes of high mortality among severely burned patients. The Efferon® LPS NEO device, originally developed for sepsis, targets both primary and secondary inflammatory mediators. This technology also shows promise in burn injury, which is characterized by a complex inflammatory response. Burn trauma triggers the release of cytokines and damage-associated molecular patterns (DAMPs), while increased intestinal permeability and endotoxin translocation may introduce pathogen-associated molecular patterns (PAMPs). Addressing both DAMPs and PAMPs is therefore critical for effective burn injury management. The goal of the study is to identify criteria for evaluating the effectiveness of hemoadsorption with the Efferon LPS NEO device in pediatric burn injury

ELIGIBILITY:
Inclusion Criteria:

* Thermal burn of Ⅱ and Ⅲ severity with a lesion area of 40% or more (ICD-10: T20-T25, T29)
* Frank index >90 (Frank Index quantifies burn severity based on the depth and total surface area of the skin lesion)
* Start of hemoadsorption no later than 5 days after admission to the ICU
* The patient should receive adequate infusion therapy (at least 30 mL/kg) from the moment of inclusion in the study until the first sorption
* The patient's condition allows Efferon LPS NEO therapy to be performed for at least 6 hours

Exclusion Criteria:

* Presence of end-stage renal disease
* Acute pulmonary embolism, confirmed by CT scan
* Uncontrolled bleeding (acute blood loss within the last 24 hours)

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with thermal burns undergoing treatment in Children's City Clinical Hospital No. 9 named after G.N. Speransky and Children's municipal multi-specialty clinical center of high medical technology
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
ICU length of stay | 1-28 days
  Time (days) from the start of hemoadsorption to transfer from the ICU

SECONDARY OUTCOMES:
Effect of the Efferon LPS NEO hemoadsoption on need for vasopressor support | 1-28 days
  Need for vasopressors according to the VIS 2020 heart rate scale (Vasoactive inotropic score)
Effect of the Efferon LPS NEO hemoadsoption on pulmonary oxygen metabolic function | 1-28 days
  Value of oxygenation index (Pa02 / Fi02 (Pa))
Effect of the Efferon LPS NEO hemoadsoption on cummulative fluid balance | 1-28 days
  Cummulative fluid balance in mL/kg
Effect of the Efferon LPS NEO hemoadsoption on duration of renal replacement therapy (RRT) | 1-28 days
  Duration of renal replacement therapy (RRT) in hours
Effect of the Efferon LPS NEO hemoadsoption on frequency of surgical interventions | 1-28 days
  Frequency of surgical interventions (necrectomy)
Effect of the Efferon LPS NEO hemoadsoption on 28 days mortality | 1-28 days
  Mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Afukov, PhD, MD, Principal Investigator — Filatov Children's City Clinical Hospital of the Moscow Health Department
Locations (2):
- Russia (2):
  - Children's City Clinical Hospital No. 9 named after G.N. Speransky of the Moscow City Health Department, Moscow
  - Children's municipal multi-specialty clinical center of high medical technology, Saint Petersburg